CLINICAL TRIAL: NCT06146907
Title: A Comparison Between the Effect of Cognitive-Motor Dual-Task Exercise Program and Exergaming on Balance, Functional Mobility, and Executive Function Among Children With Down Syndrome: A Randomized Comparative Trail
Brief Title: A Comparison of Cognitive-Motor Dual-Task Exercise and Exergaming on Balance, Functional Mobility, and Executive Function in Down Syndrome Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: safia Darweesh halwsh (Other)
Responsible Party: Sponsor-Investigator, safia Darweesh halwsh, Principal Investigator, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: exergaming and CMDT
Record Dates: First submitted 2023-11-07; First posted 2023-11-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the assessor will be blind to the allocation of participants in the two groups. the participants will not be aware of the presence of other treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive motor dual task (Active Comparator): 24 participants
  Interventions: Other: cognitive motor dual task exercises
- exergaming (Active Comparator): 24 participants
  Interventions: Other: exergaming

INTERVENTIONS:
Other: cognitive motor dual task exercises — exercise program that combined motor tasks such as walking and juggling with cognitive task such as naming fruits or colors in the room.
  Arms: cognitive motor dual task
Other: exergaming — Nintendo switch games that involve physical activity by participants to complete
  Arms: exergaming

SUMMARY:
Down syndrome (DS) is a genetic condition that compromises physical and cognitive function. Motor development delays define DS. Additionally, there are executive function issues. Humans need dual-task activities to execute physical and cognitive tasks simultaneously. Cognitively challenged people may struggle to do dual tasks simultaneously. This shows that executive function modulation may boost motor function. Rehabilitation should include motor training and cognitive therapy to improve function. Dual-task training called exergaming combines video games with exercise and requires brain processing, decision-making, and problem-solving. Kids enjoy therapy and exercise using interactive exergames, improving adherence and results. Mental agility can be developed through simultaneous exercise. Exergaming improves balance, functional mobility, fitness, and well-being for DS youngsters. Most literature on DS children stresses physical ability over cognitive ability. Cognitive-Motor Dual-Task Exercise Program (CMDT) works in most therapy settings without equipment. Our study compares two dual-task intervention regimens for 8-14-year-old DS children's balance, functional mobility, and EF.

DETAILED DESCRIPTION:
An extra copy of chromosome 21 causes Down syndrome (DS), a hereditary disorder that affects physical and cognitive function. Motor development delays characterize DS. Muscle weakness, hypotonia, and joint laxity cause motor delay. DS children demonstrated lower cognitive and motor performance in all categories than their chronological or mental-age peers. Physical traits cause DS children to struggle with balance, coordination, and functional mobility. Additionally, these kids may have executive function difficulties. Executive function helps people plan, organize, problem-solve, and control their behavior. Executive dysfunction affects impulse control, memory, attention, and decision-making. Executive and motor function are linked in several studies. Motor coordination and regulation need inhibition, working memory, and cognitive flexibility. Inhibitory control helps people stop unimportant motions for better motor skills. Working memory stores and manipulates motor plans, improving complex action execution. Motor skills affect cognitive flexibility, or the ability to alter tasks or conceptual groups. DS children show moderate inhibitory control and task initiation but poor working memory, monitoring, planning, organizing, and cognitive flexibility. Most abilities stayed consistent from 2 to 18 years. Motor and cognitive skill interventions may help DS youngsters realize their potential. EF improves with training. The dual-task physical therapy rehabilitation strategy is well studied. Living requires DT because it lets individuals perform physical and cognitive tasks simultaneously. Soccer and basketball involve coordination of motor (running, passing, and shooting) and cognitive (strategic thinking, decision-making, situation awareness) skills. DT tasks can be difficult to execute simultaneously, especially for cognitively impaired people. DT and multitasking abilities are needed. This suggests EF modulation may improve motor function. To increase function, rehabilitation programs should include motor training and cognitive therapy. Little is known about organizing physical and cognitive skill intervention programs. Exergaming is DT training that blends video games with exercise, requires mental processing, decision-making, and problem-solving. Interactive exergames make treatment and exercise more fun for kids, enhancing adherence and results. Mental agility can be increased by exercising simultaneously. DS kids can improve balance, functional mobility, fitness, and well-being through exergaming. Even so, most literature on DS children emphasizes physical capabilities over cognitive capabilities. The Cognitive-Motor Dual-Task Exercise Program (CMDT) by is a new, simple intervention that works in most therapy settings without equipment. Children's balance and movement improve with DS. The program involves walking, sitting, leaping, cognitive exercises like naming fruits and vegetables, and motor ones like carrying an empty box. our study aim to compare two DT intervention regimens for 8-14-year-old DS children's balance, functional mobility, and EF.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Down syndrome who are 8 to 14 years old.
2. Mild mental retardation (IQ according to the intelligence scale, mild (IQ 50-70).
3. Can stand and walk independently.
4. Follow verbal directions.

Exclusion Criteria:

1. Uncontrollable medical disorders or seizures.
2. Any type of disability that limits activity, such as spinal deformity.
3. Uncooperative or cannot follow instructions.
4. Children who play video games on a regular basis to avoid the extraneous activity learning effect.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of the cognitive-motor dual-task training on balance. | 6 weeks
  investigators will use Four-Square Step Test, which measures in seconds and will be compared to normative data for Down syndrome children
To investigate the effect of Cognitive Motor Dual Task training on functional mobility | 6 weeks
  investigators will use the Timed Up and Go test (measured in seconds) and compare the results for each child as pre- and post-intervention, with less time indicating improvements.
To investigate the effect of the exergaming training on balance. | 6 weeks.
  investigators will use Four-Square Step Test, which measures in seconds and will be compared to normative data for Down syndrome children
To investigate the effect of exergaming training on functional mobility | 6 weeks
  investigators will use the Timed Up and Go test (measured in seconds) and compare the results for each child as pre- and post-intervention, with less time indicating improvements.
To investigate the effect of the cognitive-motor dual-task training on balance. | 6 weeks
  investigators will use Pediatric Balance Scale (Maximum score = 56 points, with 56 points being a perfect score)
To investigate the effect of the exergaming training on balance. | 6 weeks
  investigators will use Pediatric Balance Scale (maximum score = 56 points, with 56 points being a perfect score).

SECONDARY OUTCOMES:
To examine the effect of cognitive-motor Motor Dual Task on Executive Function | 6 weeks
  investigators will use the Cambridge Neuropsychological Test Automated Battery (measured in seconds; less time to complete the test indicates improvement).
To examine the effect of exergaming on Executive Function | 6 weeks
  investigators will use the Cambridge Neuropsychological Test Automated Battery (measured in seconds; less time to complete the test indicates improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
This study's individual participant data (IPD) will be shared in conformity with Saudi Arabian law, PNU/IRB policy, and ICH Good Clinical Practice recommendations. IPD will include study protocol and statistics analysis plan. With PNU/IRB permission and a data sharing agreement, we will make the IPD available to other researchers upon request. To request IPD, contact the investigator with the subject line "Request for IPD from [study title]." Within a year following the primary study results, we will provide the IPD. IPD requests beyond this period will be examined individually. We will not disclose IPD with participant names, addresses, or contact information. We will protect the IPD according to PNU/IRB policies and ICH Good Clinical Practice recommendations. The IPD will be securely stored and only authorized personnel can access it.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after publication
Access Criteria: The researcher is affiliated with a recognized academic or research institution.
  The researcher has a clear and well-defined research proposal that is relevant to the study and aims to generate new knowledge or insights.
  The researcher has the necessary expertise and resources to analyze the IPD and generate meaningful results.
  The researcher agrees to comply with all relevant rules and regulations, including those related to data privacy and confidentiality.
  The researcher agrees to use the IPD solely for the purpose of the approved research proposal and not for any commercial or other purposes.
  The researcher agrees to provide regular updates on the progress of the research and to share any resulting publications or findings with the study team.
  The researcher agrees to comply with any additional requirements or conditions set by the study team or the data provider.

REFERENCES:
- [Derived] Halwsh SD, Algabbani MF, Alqabbani S, Alahmad TA, Almurdi MM, Alshubaily RA, Aldera M, Al-Dubisi HA, Almedlej RM, Shaheen AAM. The Effects of Cognitive-Motor Dual-Task Exercise and Exergaming on Balance and Functional Mobility in Children with Down Syndrome: A Comparative Randomized Trial. Brain Sci. 2026 Jan 6;16(1):79. doi: 10.3390/brainsci16010079. PMID 41594800